CLINICAL TRIAL: NCT04771494
Title: Effect of Instability on Power and Speed in Bench Press
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, Moisés Marquina Nieto, Principal Investigator, Universidad Politecnica de Madrid
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Power and speed in instability
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Instability, Joint
Keywords: Strength Training; Unstable Devices; Balance; Speed Training; Core
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trained (Experimental): Participants with at least 6 months of training with unstable devices
  Interventions: Other: Power and execution speed as a function of instability experience
- Untrained (Experimental): Participants with no previous instability experience
  Interventions: Other: Power and execution speed as a function of instability experience

INTERVENTIONS:
Other: Power and execution speed as a function of instability experience — Each subject performed 3 repetitions for the light load (40% RM; VMP > 1.0 m/s), with 1 minute rest; 2 repetitions for the medium load (60% RM; 0.65 m/s ≤ VMP ≤ 1.0 m/s) with 2 minutes rest and 1 repetition for the heavy load (80% RM; VMP < 0.65 m/s) with 4 minutes rest. A metronome was used for the start countdown and to time the eccentric and concentric portions of the exercise.
  Subjects began the bench press with their elbows fully extended, maintaining a grip distance slightly greater than shoulder width. The bar was then lowered to their chest and then applying as much thrust as possible until full elbow extension on a 2-1-0 count. The timing sequence involved 2 seconds for the eccentric phase, a 1 second hold (to minimise the contribution of the rebound effect and allow for more reproducible and consistent measurements) and for the concentric "up" phase the highest possible execution speed, until the bar returned to the starting position.

SUMMARY:
The aim of this study was to analyse and compare the speed and power parameters in bench press training in different degrees of instability: 1) stable (PBE), 2) with asymmetric load (PBA), 3) with oscillating load (PBO), 4) on fitball (PBF) and 5) on bosu (PBB). For this purpose, 20 male subjects (10 trained and 10 untrained) with specific experience in training under unstable conditions were evaluated with respect to mean propulsive velocity (MPV), maximum velocity (MV) and power (POT) with different types of external load: low load (40% of 1RM), medium load (60% of 1RM) and high load (80% of 1RM) in each condition.

DETAILED DESCRIPTION:
Therefore, the aim of this study was to analyse the effect of different degrees of instability on power and speed of execution in the bench press exercise. For the design of this quasi-experimental research, with an ad hoc protocol, an intersubject comparison was used in 5 different conditions. 20 male participants were grouped into two groups based on their previous experience with unstable training and volunteered for this study. Expert group (n= 10; 23.70 ± 4.30 years; 81.40 ± 9.67 kg; 179.50 ± 8.95 cm; 3.5 ± 4.10 years of strength training experience; 9 ± 10.60 months of unstable training experience) Novice group (n= 10; 25.60 ± 6.50 years; 77.80 ± 4.44 kg; 176.40 ± 2.80 cm; 3.40 ± 1.96 years of strength training experience; 0.90 ± 0.99 months of unstable training experience). Subjects with no experience in training with unstable loads (having implemented unstable loads in their training at some point) or current or recent injuries (within the last 6 months) that caused them to alter their normal physical activity were excluded from this study. This study was in accordance with the Declaration of Helsinki (2013). All participants gave written informed consent prior to the study.

Subjects performed the bench press exercise by assessing mean propulsive velocity and power with 3 different loads for each of the unstable situations: light (40% of 1RM), moderate (60% of 1RM) and high (80% of 1RM). In a familiarisation session, subjects performed the relative loads with each condition to determine their strength-velocity profiles and their optimal work percentages. In addition, an incremental load test was performed to determine the 1RM of each of the participants to determine the external load for each load percentage in each of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* two years of continuous strength training experience
* a minimum of 6 months of suspended training experience

Exclusion Criteria:

* Athletes who presented pain or skeletal or neuromuscular disorder

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-05-17 (Actual)

PRIMARY OUTCOMES:
Power | 1 month
  the ability to perform different actions, developing maximum strength in a short time
Maximum Speed | 1 month
  maximum value of m/s reached during the exercise
Mean Propulsive Speed | 1 month
  the average speed reached during the concentric phase of the exercise is recorded

CONTACTS AND LOCATIONS:
Overall Officials: Moisés M Marquina Nieto, Principal Investigator — Univerdidad Politécnica de Madrid
Locations (1):
- Facultad Ciencias de la Actividad Física y del Deporte, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No